CLINICAL TRIAL: NCT00173342
Title: Congenital or Idiopathic Complete Right Bundle Branch Block: Physiological Significance and Molecular Characterization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700620
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Bundle-Branch Block
Keywords: Right bundle branch block; Electrocardiography; Ion channel
MeSH Terms: conditions — Bundle-Branch Block

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
This study is to determine 1) the incidence of altered right bundle conduction, including CRBBB, IRBBB or rsR' pattern in the Taipei city based on the school survey databank from 1999 to 2002, 2) the associated cardiac lesions, 3) clinical presentations relevant to the altered right bundle conduction, 4) the association with QTc prolongation and dispersion and HRV from a 5-minutes recording. Finally, molecular characterization for those with CRBBB or Brugada pattern EKG, especially those with positive family history will be studied.

DETAILED DESCRIPTION:
The EKG pattern and medical records from the school survey from 1999 to 2002 in Taipei city will be reviewed, and the basic data of those with CRBBB, IRBBB and rsR' pattern will be recorded. Interview will be made and the echocardiographic measurements will be performed to identify associated cardiac defects. EKG parameters and QT, QTc, QT dispersion, QTc dispersion and HRV parameters will be obtained from a semi-automated system. Time domain and frequency domain measures will be calculated and expressed as SDNN, triangular index, SDNN index, total power, low frequency power and high frequency power. Mutational analysis and DNA sequencing will be conducted in those with CRBBB or Brugada pattern EKG, especially those with positive family history.

Based on these data, the clinical significance of altered bundle branch conduction identified from a school survey may be defined. For those with isolated CRBBB or IRBBB, the adjunctive value of HRV and QT parameters will determined the high risk group, and 24 hour Holter recording and Treadmill exercise test will then perform in these patients to define association with ventricular arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* ECG showed right bundle branch block

Exclusion Criteria:

* can't tolerate Treadmill ECG study

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hwan Wu, MD, PhD, Study Chair — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - Department of Pediatrics, National Taiwan University Hospital, Taipei
  - Pediatric Department, National Taiwan University Hospital, Taipei